CLINICAL TRIAL: NCT01519648
Title: A Russian Prospective Observational Study of Invasive Fungal Infections in Patients With Acute Leukemia and Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: National Hematological Society, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: RIFI
Record Dates: First submitted 2012-01-23; First posted 2012-01-27 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Invasive Fungal Infections
Keywords: Invasive fungal infection; Acute leukemia (AL); Hematopoietic stem cell transplantation; Antifungal stewardship; Neutropenia; Hematological malignancies
MeSH Terms: conditions — Invasive Fungal Infections; Neutropenia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute leukemia patients: Patients with de novo or relapsed acute myeloid and lymphoid leukemia
- Allo- or auto- transplant recipients

SUMMARY:
Estimate the rate of occurrence of Invasive Fungal Infections (IFIs) in patients with acute leukemia for the first 6 months of chemotherapy (that usually correspond to four courses of chemotherapy), and hematopoietic stem cells transplantation.

DETAILED DESCRIPTION:
This multi-center observational study of IFI in high risk hematological patients, the study will investigate the epidemiology of IFI, describe antifungal strategy, proportion of antifungal prophylaxis, empiric therapy, pre-emptive therapy and targeted therapy in at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with de novo or relapsed AL (AML, ALL)started chemotherapy
* All newly allogeneic or autologous transplant recipients during the study period

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational study will be implemented in the hematology departments or hematology centers with or without HSCT located throughout Russia.
Sampling Method: Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galina A Klyasova, Principal Investigator — National Research Center for Hematology
Locations (1):
- National Hematological Society, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Leukemia Patients | Allo- or Auto- Transplant Recipients
Started | 502 | 306
Completed | 502 | 306
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Leukemia Patients | Allo- or Auto- Transplant Recipients | Total
Number analyzed (Participants) | 502 | 306 | 808
Age, Continuous [Median (Full Range); unit: years] | 42 (1-79) [1 to 79] | 37 (1-66) [1 to 66] | 40 (1-79) [1 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 69 | 55 | 124
  Between 18 and 65 years | 389 | 250 | 639
  >=65 years | 44 | 1 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 261 | 150 | 411
  Male | 241 | 156 | 397
Region of Enrollment [Number; unit: participants]
  Russian Federation | 502 | 306 | 808

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Invasive Fungal Infections
Description: Estimate the rate of IFIs in patients with acute leukemia for the first 6 months of chemotherapy (that usually correspond to four courses of chemotherapy), and hematopoietic stem cells transplantation.
Time Frame: 6 month
Measure: Number; unit: participants
Groups:
- Allo- or Auto- Transplant Recipients: Allo- or auto- transplant recipients
Arm/Group | Acute Leukemia Patients | Allo- or Auto- Transplant Recipients
Number analyzed (Participants) | 502 | 306
participants | 77 | 27
Statistical Analysis 1: Comparison: Acute Leukemia Patients vs Allo- or Auto- Transplant Recipients; Test type: Superiority or Other; p = 0.007, Chi-squared; Odds Ratio (OR) = 1.872, 95% CI 2-sided [1.178 to 2.977], Standard Error of Mean 0.237

ADVERSE EVENTS:
Description: The study was observational and the adverse events were not evaluated
Arm/Group | Acute Leukemia Patients | Allo- or Auto- Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No